CLINICAL TRIAL: NCT03956719
Title: Efficacy and Safety of Autologous Adipose-derived Mesenchymal Stem Cells in the Treatment of Early Knee Osteoarthritis
Brief Title: Treatment of Early Knee Osteoarthritis With Autologous Adipose-derived Mesenchymal Stem Cells
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019042
Record Dates: First submitted 2019-05-16; First posted 2019-05-21 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Knee Osteoarthritis
Keywords: Autologous adipose-derived mesenchymal stem cells; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous adipose-derived mesenchymal stem cells (Experimental): Patients receiving intra-articular injection of autologous adipose-derived mesenchymal stem cells
  Interventions: Drug: Autologous adipose-derived mesenchymal stem cells; Procedure: abdominal liposuction

INTERVENTIONS:
Drug: Autologous adipose-derived mesenchymal stem cells — Autologous adipose-derived mesenchymal stem cells is extracted from human abdominal fat, which is crushed, filtered and immediately returned to the articular cavity through a specific device.
Procedure: abdominal liposuction — 50 ml abdominal fat was extracted by abdominal liposuction to prepare autologous adipose-derived mesenchymal stem cells

SUMMARY:
The purpose of this study is to explore the efficacy and safety of autologous adipose mesenchymal stem cells in the treatment of early knee arthritis. Investigator believes that autologous adipose mesenchymal stem cells can relieve pain, improve knee function, promote knee cartilage regeneration and improve life satisfaction of patients.

DETAILED DESCRIPTION:
Investigators extracted abdominal fat from eight patients, extracted autologous adipose mesenchymal stem cells and injected them into the knee joint of the patients. The data were followed up regularly after operation and compared with those before operation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years, male and female, patient can tolerate surgery;
* Clinical diagnosis of early stage degenerative arthritis by Radiographic Criteria and physical examination;
* Obviously extra-articular malformation;
* Course of disease ≥ six months;
* No medication for knee osteoarthritis in the past three months
* Evaluated has not at the risk of cancer;
* Subjects who understand and sign the consent form for this study.

Exclusion Criteria:

* Acute joint injury;
* Patients with severe primary diseases, such as cardiovascular,cerebrovascular, liver, kidney and hematopoietic system, and psychosis;
* Cancer patients;
* Women who are pregnant or breast feeding,or allergic constitution patient;
* Positive serology for HIV-1 or HIV-2, Hepatitis B (HBsAg, Anti-Hepatitis C virus -Ab), Hepatitis C (Anti-hepatitis C virus -Ab) and syphilis;
* Receive other open surgery related to knee operation within 6 months;
* Participation in another clinical trial;
* Failing to comply with the inclusion criteria, unwilling to comply with the research approach, or incomplete data affecting the curative effect or safety judgment.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2019-03-02 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Hospital for special surgery knee score postoperative 1 month | postoperative 1 month
  Hospital for special surgery knee score is a knee function scoring system with a full score of 100. 0 means the loss of knee function, 100 means the best knee function, and the greater the value, the better knee function.
Hospital for special surgery knee score postoperative 3 month | postoperative 3 month
  Hospital for special surgery knee score is a knee function scoring system with a full score of 100. 0 means the loss of knee function, 100 means the best knee function, and the greater the value, the better knee function.
Hospital for special surgery knee score postoperative 6 month | postoperative 6 month
  Hospital for special surgery knee score is a knee function scoring system with a full score of 100. 0 means the loss of knee function, 100 means the best knee function, and the greater the value, the better knee function.
Visual Analogue Scale Postoperative 1 month | Postoperative 1 month
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Visual Analogue Scale Postoperative 3 month | Postoperative 3 month
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Visual Analogue Scale Postoperative 6 month | Postoperative 6 month
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Evaluation of cartilage repair under MRI postoperative 3 month | postoperative 3 month
  Recht criterion was used for grading articular cartilage injury of knee joint, including 0-IV grade, in which: 0 grade, normal articular cartilage, no obvious abnormal signal was found; 1 grade, the layered structure of cartilage disappeared, and there were focal low signal areas, but the surface was smooth; 2 grade, the surface of cartilage was irregular, the depth of cartilage injury was less than 50% cartilage thickness; 3 grade, the surface of cartilage was heavy. The degree of injury is irregular, the depth of injury is more than 50% of the thickness of cartilage or through the whole layer, but the surface of cartilage is not completely exfoliated; Grade IV, full-thickness cartilage defect, articular cartilage injury deep to the cortex, subchondral bone exposed.
Evaluation of cartilage repair under MRI postoperative 6 month | postoperative 6 month
  Recht criterion was used for grading articular cartilage injury of knee joint, including 0-IV grade, in which: 0 grade, normal articular cartilage, no obvious abnormal signal was found; 1 grade, the layered structure of cartilage disappeared, and there were focal low signal areas, but the surface was smooth; 2 grade, the surface of cartilage was irregular, the depth of cartilage injury was less than 50% cartilage thickness; 3 grade, the surface of cartilage was heavy. The degree of injury is irregular, the depth of injury is more than 50% of the thickness of cartilage or through the whole layer, but the surface of cartilage is not completely exfoliated; Grade IV, full-thickness cartilage defect, articular cartilage injury deep to the cortex, subchondral bone exposed.
Degree of meniscus injury under MRI postoperative 3 month | postoperative 3 month
  Stoller's criteria were used in the classification of meniscal injuries, including 0-3 grades, in which: 0 grade, the shape of meniscus was regular, complete and even low signal; 1 grade, focal ellipse or circular high signal appeared in the meniscus, which did not extend to the articular surface and margin of the meniscus; 2 grade, the meniscus showed horizontal linear high signal extending to the articular margin of the meniscus.
  But it did not exceed the articular surface; in grade III, the shape of meniscus was irregular and incomplete. Irregular or linear high signal appeared in the meniscus and extended to the articular surface of meniscus. The grade I and II symptoms of meniscus injury were mild, suggesting meniscus degeneration, and grade III suggesting meniscus tear.
Degree of meniscus injury under MRI postoperative 6 month | postoperative 6 month
  Stoller's criteria were used in the classification of meniscal injuries, including 0-3 grades, in which: 0 grade, the shape of meniscus was regular, complete and even low signal; 1 grade, focal ellipse or circular high signal appeared in the meniscus, which did not extend to the articular surface and margin of the meniscus; 2 grade, the meniscus showed horizontal linear high signal extending to the articular margin of the meniscus.
  But it did not exceed the articular surface; in grade III, the shape of meniscus was irregular and incomplete. Irregular or linear high signal appeared in the meniscus and extended to the articular surface of meniscus. The grade I and II symptoms of meniscus injury were mild, suggesting meniscus degeneration, and grade III suggesting meniscus tear.
Squatting to Standing Time postoperative 1 month | postoperative 1 month
  The patient squatted on the floor and then stood up completely for five consecutive times, recording the time required.
Squatting to Standing Time postoperative 3 month | postoperative 3 month
  The patient squatted on the floor and then stood up completely for five consecutive times, recording the time required.
Squatting to Standing Time postoperative 6 month | postoperative 6 month
  The patient squatted on the floor and then stood up completely for five consecutive times, recording the time required.

SECONDARY OUTCOMES:
Satisfaction of patients postoperative 1 month | postoperative 1 month
  The satisfaction degree of patients with treatment effect, full score of 10 points, 1 represents not satisfied at all, 10 represents very satisfied.
Satisfaction of patients postoperative 3 month | postoperative 3 month
  The satisfaction degree of patients with treatment effect, full score of 10 points, 1 represents not satisfied at all, 10 represents very satisfied.
Satisfaction of patients postoperative 6 month | postoperative 6 month
  The satisfaction degree of patients with treatment effect, full score of 10 points, 1 represents not satisfied at all, 10 represents very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Peilai Liu, MD, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Qilu hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
The acquisition of individual participant data needs the consent of Peilai Liu, the person in charge.

REFERENCES:
- [Background] Yu D, Xu J, Liu F, Wang X, Mao Y, Zhu Z. Subchondral bone changes and the impacts on joint pain and articular cartilage degeneration in osteoarthritis. Clin Exp Rheumatol. 2016 Sep-Oct;34(5):929-934. Epub 2016 Aug 31. PMID 27606839
- [Background] Wilusz RE, Sanchez-Adams J, Guilak F. The structure and function of the pericellular matrix of articular cartilage. Matrix Biol. 2014 Oct;39:25-32. doi: 10.1016/j.matbio.2014.08.009. Epub 2014 Aug 27. PMID 25172825
- [Background] Fodor PB, Paulseth SG. Adipose Derived Stromal Cell (ADSC) Injections for Pain Management of Osteoarthritis in the Human Knee Joint. Aesthet Surg J. 2016 Feb;36(2):229-36. doi: 10.1093/asj/sjv135. Epub 2015 Aug 3. PMID 26238455
- [Background] Awad ME, Hussein KA, Helwa I, Abdelsamid MF, Aguilar-Perez A, Mohsen I, Hunter M, Hamrick MW, Isales CM, Elsalanty M, Hill WD, Fulzele S. Meta-Analysis and Evidence Base for the Efficacy of Autologous Bone Marrow Mesenchymal Stem Cells in Knee Cartilage Repair: Methodological Guidelines and Quality Assessment. Stem Cells Int. 2019 Apr 7;2019:3826054. doi: 10.1155/2019/3826054. eCollection 2019. PMID 31089328
- [Background] Senn-Malashonak A, Wallek S, Schmidt K, Rosenhagen A, Vogt L, Bader P, Banzer W. Psychophysical effects of an exercise therapy during pediatric stem cell transplantation: a randomized controlled trial. Bone Marrow Transplant. 2019 Nov;54(11):1827-1835. doi: 10.1038/s41409-019-0535-z. Epub 2019 May 14. PMID 31089282
- [Background] Browne JA, Nho SJ, Goodman SB, Callaghan JJ, Della Valle CJ. Stem Cells and Platelet-Rich Plasma Injections for Advanced Hip and Knee Arthritis: Enthusiasm Outpaces Science. J Arthroplasty. 2019 Jun;34(6):1049-1050. doi: 10.1016/j.arth.2019.03.074. Epub 2019 Apr 3. No abstract available. PMID 31000403
- [Background] Strotman PK, Novicoff WM, Nelson SJ, Browne JA. Increasing Public Interest in Stem Cell Injections for Osteoarthritis of the Hip and Knee: A Google Trends Analysis. J Arthroplasty. 2019 Jun;34(6):1053-1057. doi: 10.1016/j.arth.2019.03.002. Epub 2019 Mar 8. PMID 30935801
- [Background] Chareancholvanich K, Pornrattanamaneewong C, Narkbunnam R. Increased cartilage volume after injection of hyaluronic acid in osteoarthritis knee patients who underwent high tibial osteotomy. Knee Surg Sports Traumatol Arthrosc. 2014 Jun;22(6):1415-23. doi: 10.1007/s00167-013-2735-1. Epub 2013 Oct 27. PMID 24162762